CLINICAL TRIAL: NCT07278583
Title: Eligibility Criteria Evaluation of Heart Failure Telemonitoring : Analysis of CARDIAUVERGNE's Cohort
Brief Title: Evaluation of Heart Failure Telemonitoring Eligibility Criteria
Acronym: Weigh-HF
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2025 RIOCREUX
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
Keywords: heart failure; telemonitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to analyze the prognosis and evolution of patients after exclusion of CARDIAUVERGNE, a heart failure telemonitoring system at Clermont-Ferrand's hospital. The patients were included from 1st January 2023 to 31st December 2024 and the monitoring was terminated for end of eligibility according to the french health authority criteria.

DETAILED DESCRIPTION:
After an episode of heart failure, patients have been included in a telemonitoring program in order to reduce rehospitalizations for heart failure and improve follow-up. On a daily basis, the patients weigh themselves on connected scales which enables a team of dedicated nurses to follow them closely. If need be they can call the patient, ask for a blood exam and adapt their prescription. Indeed, if remote support is insufficient, patients can be hospitalized prematurely and so decrease the duration of hospital care.

The inclusion criteria correspond to either an episode of heart failure in the last 12 months or dyspnea at least NYHA2 with NT-proBNP over 1000pg/mL.

The follow up is renewed every 6 months. Patients are excluded from monitoring when criteria are no longer fulfilled. As these characteristics have been chosen empirically, our aim is to see if patients no longer presenting these standards have indeed a low chance of bad evolution.

Information is gathered from their medical record at inclusion, exclusion and 1 year after exclusion. A short phone call is made after 1 year of exclusion, to appreciate their evolution and gather information concerning their symptoms, treatments ...

ELIGIBILITY:
Inclusion Criteria:

* adults
* able to read and understand french
* included in CARDIAUVERGNE telemonitoring program from 1st january 2023 to 31st december 2024 such as defined by the french health authorithy criteria (heart failure within 12 months or dyspnea at least NYHA 2 associated with NTproBNP of at least 1000pg/mL) and excluded by medical decision as no longer presenting eligibillity criteria

Exclusion Criteria:

* Patients leaving telemonitoring for other reasons (choice, death, medical reason, relocation, inobservance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in CARDIAUVERGNE telemonitoring that have been excluded as they no longer fulfill the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite criterion defined by the occurrence within one year following the end of remote monitoring of either cardiovascular death or heart failure worsening (hospitalization or unscheduled visit for heart failure) | From telemonitoring exclusion up to a year after

SECONDARY OUTCOMES:
Amount of medical appointments | From telemonitoring exclusion up to a year after
  General practician and cardiology consultations
Natriuretic peptides evolution | From inclusion until a year after exclusion
  Comparison at inclusion, exclusion and a year after exclusion for monitoring
Amount of theoretically possible re-included patients during follow up | From telemonitoring exclusion up to a year after
Determination of potential patient profiles more suitable to discontinue remote monitoring | From inclusion up to a year after telemonitoring exclusion

CONTACTS AND LOCATIONS:
Overall Officials: Clément RIOCREUX, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savarese G, Lund LH. Global Public Health Burden of Heart Failure. Card Fail Rev. 2017 Apr;3(1):7-11. doi: 10.15420/cfr.2016:25:2. PMID 28785469
- [Background] Rapport au parlement "évaluation des expérimentations de télésurveillance du programme national étapes" Novembre 2020
- [Background] Haute Autorité Santé. "Télésurveillance médicale du patient insuffisant cardiaque chronique," 2023.
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2022 Jan;24(1):4-131. doi: 10.1002/ejhf.2333. PMID 35083827